CLINICAL TRIAL: NCT06098053
Title: Efficacy of Muscle Energy Technique Alone and in Combination With Interferential Therapy for the Treatment of Non-specific Low Back Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuro Counsel Hospital, Pakistan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 348
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Intervention Model Description: Single blind RCT in which Two groups were formed
Who Masked: Participant
Masking Description: Just participants were unaware of which intervention they are being given
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Muscle energy technique was given to this group
  Interventions: Other: muscle energy technique
- Group B (Active Comparator): Muscle energy technique along with interferential therapy was given to this group
  Interventions: Other: Muscel energy technique along with interferential therapy

INTERVENTIONS:
Other: muscle energy technique — Muscle energy technique is used at a rate of three sessions per week for four and half weeks
  Arms: Group A
Other: Muscel energy technique along with interferential therapy — Muscle energy technique along with interferential therapy is used at a rate of three sessions per week for four and half weeks
  Arms: Group B

SUMMARY:
Single blind randomized control trail in which two groups were formed. Group A was given Muscle energy technique and Group B was given muscle energy technique in combination with Interferential therapy.

DETAILED DESCRIPTION:
After getting the REC approval from The Neurocounsel Clinics, study was initiated from 21 May, 2023 to 20 September 2023. Sample size was calculated by Epitool which came 30. Following participants were included a) both genders b) age 20-50 years and followings were excluded a) DM b) Parkinson disease c) disc disorder d) MSK disorder were excluded from this study. Simple random sampling technique was used to randomize participants into two equal groups. group A was given MET and group B was given MET plus IFT. 2 sessions/week for 4 & half weeks. Evaluation was done at PNS & EQ-5D-5L (QoL). Pre and post test analysis was done by use of SPSS version 21 and level of significance was kept p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* both genders
* age between 20-50 years old
* non specific type of back pain

Exclusion Criteria:

* Diabetes Mellitus
* Parkinson disease
* Any other Musculoskeletal disorder

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-21 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Pain numeric scale | 4 and half weeks
  this scale is used to measure the pain 0 means no pain and 10 means worst pain ever
short form of 36 | 4 and half weeks
  SF-36 is used to meaure the quality of life. 0 means worst quality of life and higher values towards 100 means best quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- The Neurocouncil Clinic, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
have not decided anything yet